CLINICAL TRIAL: NCT03206255
Title: Immuno-persistence Study of A Bivalent Human Papillomavirus (Type 16, 18) Recombinant Vaccine (E.Coli) in Healthy Female Subjects Aged 9 to 17 Years
Brief Title: Immuno-persistence Study of a Recombinant Human Papillomavirus 16/18 Bivalent Vaccine in Preadolescent Girls
Status: Completed | Type: Observational
Sponsor: Jun Zhang (Other)
Collaborators: Xiamen Innovax Biotech Co., Ltd (Industry); Beijing Wantai Biological Pharmacy Enterprise Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Jun Zhang, Professor, Xiamen University
Organization: Xiamen University (Other)
Other Study IDs: HPV-PRO-006-2
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Cancer; Vaginal Intraepithelial Neoplasia; Vulvar Intraepithelial Neoplasia; Persistent Infection
Keywords: Human Papilloma Virus 16; Human Papilloma Virus 18; adolescent girl; non-inferiority; immuno-persistence
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms; Persistent Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 9-17y (0,1,6m): Participants in this arm have received 60μg of HPV 16/18 bivalent vaccine according to 3 doses of HPV 16/18 bivalent vaccine
  Interventions: Procedure: 3 doses of HPV 16/18 bivalent vaccine
- 9-14y (0,6m): Participants in this arm have received 60μg of HPV 16/18 bivalent vaccine according to 2 doses of HPV 16/18 bivalent vaccine
  Interventions: Procedure: 2 doses of HPV 16/18 bivalent vaccine
- 18-26y (0,1,6m): Participants in this arm have received 60μg of HPV 16/18 bivalent vaccine according to 3 doses of HPV 16/18 bivalent vaccine
  Interventions: Procedure: 3 doses of HPV 16/18 bivalent vaccine

INTERVENTIONS:
Procedure: 3 doses of HPV 16/18 bivalent vaccine — Participants have received 60μg of HPV 16/18 bivalent vaccine according to the standard 3-dose schedule (0,1,6 months)
  Groups: 18-26y (0,1,6m); 9-17y (0,1,6m)
Procedure: 2 doses of HPV 16/18 bivalent vaccine — Participants have received 60μg of HPV 16/18 bivalent vaccine according to an alternative 2-dose schedule (0,6 months)
  Groups: 9-14y (0,6m)

SUMMARY:
The primary objective of this study is to evaluate the immuno-persistence (type specific IgG antibody) of the tested vaccine administered in girls aged 9-17 years ,comparing to young healthy adults of 18-26 years who received the standard 3-dose schedule (0,1,6 months).

DETAILED DESCRIPTION:
This is a follow-up study which is based on the bridging study of a recombinant human papillomavirus 16/18 bivalent vaccine in preadolescent girls(Unique Protocol ID:HPV-PRO-006,Identifiers: NCT02562508) .We will recruit people who have participated in bridging study before and collect their serum samples to test the seroprevalence and geometric mean concentrations of anti-HPV16 and anti-HPV18 antibody on 18 and 30 months after dose 1.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who participated in the bridging study of a recombinant human papillomavirus 16/18 bivalent vaccine in preadolescent girls (Unique Protocol ID:HPV-PRO-006-2, Identifiers: NCT02562508) and received at least one dose;
2. The legal guardian of participants under age 18 can provide identity certificate, or representative can provide authorization;
3. Participants under the age 18, able to sign or whose legal guardian agree to sign the written informed consent; or participants aged 18 and older agree to sign the written informed consent;
4. Able to comply with the requests of the study;

Exclusion Criteria:

1. Participants with coagulation dysfunction (such as coagulation factor deficiency, blood-clotting disorder, or platelet disorder) or coagulation disorders, as diagnosed by a physician after vaccination ;
2. According to the investigator's judgment, there might be some medical, psychological, social or occupational factors which might impact on the individual to obey the protocol or sign the informed consent;

Ages: 10 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants who participated in the bridging study (Unique Protocol ID:HPV-PRO-006-2, Identifiers: NCT02562508) and received at least one dose will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 940 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Anti-HPV16 and anti-HPV18 seroprevalence and geometric mean concentrations at Months 18 and 30 (type specific IgG antibody) | Month 18 and 30
  To detect the anti-HPV 16 and anti-HPV 18 type specific IgG antibody level on 18 and 30 months after the dose 1

SECONDARY OUTCOMES:
Anti-HPV16 and anti-HPV18 seroprevalence and geometric mean concentrations at Months 18 and 30 (type specific neutralizing antibody) | Month 18 and 30
  To detect the anti-HPV 16 and anti-HPV 18 type specific neutralizing antibody level on 18 and 30 months after the dose 1
All the Serious Adverse Events(SAE) occurred during clinical trial time frame would be recorded | between 7 months and 30months after the dose1

CONTACTS AND LOCATIONS:
Overall Officials: Ting Wu, Ph. D., Study Chair — Xiamen University; Yuemei Hu, Bachelor, Principal Investigator — Jiangsu Provincial Centre for Disease Control and Prevention
Locations (1):
- Jiangsu Provincial Centre for Disease Control and Prevention, Nanjing, Jiangsu, China